CLINICAL TRIAL: NCT06187792
Title: Constructing a Model of Pupillary Parameters in Predicting Delirium Among Critically Ill Patients in the Intensive Unit
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: National Taiwan University Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: 202306099DINA
Record Dates: First submitted 2023-12-17; First posted 2024-01-03 (Actual); Last update posted 2024-01-03 (Actual); Status verified 2023-10

CONDITIONS: ICU Delirium
Keywords: Delirium; Predicting delirium; Automated Infrared Pupillometry (AIP); Pupil Parameters; Intensive Care Delirium Screening Checklist (ICDSC)
MeSH Terms: conditions — Delirium

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Delirium is commonly observed in critically ill patients in intensive care units (ICUs), imposing significant burdens on both patients and the healthcare system. Existing assessment tools have certain limitations. Studies have indicated a correlation between pupil parameters and neurological disorders including delirium. Automated Infrared Pupillometry, widely used in neurological disorders, is employed in this study to assess its accuracy and predictive power in evaluating delirium among critically ill patients. The aim is to investigate the accuracy and predictive capability of these parameters in assessing delirium, while identifying the optimal cut-off points. The research findings will contribute to enhancing early detection and prevention of delirium in ICU settings.

DETAILED DESCRIPTION:
Delirium is an acute impairment of attention and cognitive function commonly observed in critically ill patients in intensive care units (ICUs). It leads to long-term cognitive impairment and increased risk of mortality for patients, while also causing distress for healthcare providers and family members, imposing substantial burdens on patients, families, and healthcare systems. Although there are assessment tools and predictive models available for detecting delirium, they have certain limitations.

Recent studies have indicated an association between delirium and the neurotransmitter acetylcholine (ACh). Acetylcholine not only regulates consciousness and cognitive wakefulness but also modulates pupil constriction and light reflex. In clinical practice, the Automated Infrared Pupillometry (AIP) has emerged as a robust tool for assessing acetylcholine, aiding in early delirium detection. However, more research is needed to clearly establish their relationship. This study aims to investigate the accuracy and predictive power of Automated Infrared Pupillometry in assessing delirium among critically ill patients. It involves collecting pupil parameters from critically ill patients and examining the correlation between delirium and pupil parameters using the Intensive Care Delirium Screening Checklist (ICDSC). The goal is to explore the accuracy and predictive capability of these parameters in evaluating delirium, identifying optimal cut-off points. The findings will contribute to enhancing early detection and prevention of delirium in intensive care settings.

ELIGIBILITY:
Inclusion Criteria:

* Patients admitted to the intensive care unit from internal and surgical departments.
* Ages 18 and above.

Exclusion Criteria:

* Acute brain injury (hemorrhagic, ischemic stroke).
* Other brain-related diseases (brain tumor, brain infection, oculomotor nerve paralysis, etc.).
* Ophthalmic diseases that prevent monitoring of pupil measurements.
* Patients with pre-hospital cardiac arrest or in-hospital cardiac arrest.
* Estimated stay in the intensive care unit not exceeding 72 hours.
* Refusal to participate in this study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients admitted to the intensive care unit from internal and surgical departments.
Sampling Method: Non-Probability Sample
Enrollment: 200 (Estimated)
Dates: Start 2023-10-04 (Actual); Primary Completion 2025-09 (Estimated); Study Completion 2025-09 (Estimated)

PRIMARY OUTCOMES:
Constructing a model based on pupillary parameters and delirium: | 2023/09/1-2025/08/30
  By analyzing the relationship between pupillary parameters and delirium, identifying the optimal cut-off point, and constructing a formula.

CONTACTS AND LOCATIONS:
Locations (1):
- Ming-Chen Chiang, Taipei, Taiwan

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Almeida IC, Soares M, Bozza FA, Shinotsuka CR, Bujokas R, Souza-Dantas VC, Ely EW, Salluh JI. The impact of acute brain dysfunction in the outcomes of mechanically ventilated cancer patients. PLoS One. 2014 Jan 22;9(1):e85332. doi: 10.1371/journal.pone.0085332. eCollection 2014. PMID 24465538
- [Result] Bergeron N, Dubois MJ, Dumont M, Dial S, Skrobik Y. Intensive Care Delirium Screening Checklist: evaluation of a new screening tool. Intensive Care Med. 2001 May;27(5):859-64. doi: 10.1007/s001340100909. PMID 11430542
- [Result] Bujang MA, Adnan TH. Requirements for Minimum Sample Size for Sensitivity and Specificity Analysis. J Clin Diagn Res. 2016 Oct;10(10):YE01-YE06. doi: 10.7860/JCDR/2016/18129.8744. Epub 2016 Oct 1. PMID 27891446
- [Result] Carnahan RM, Lund BC, Perry PJ, Pollock BG, Culp KR. The Anticholinergic Drug Scale as a measure of drug-related anticholinergic burden: associations with serum anticholinergic activity. J Clin Pharmacol. 2006 Dec;46(12):1481-6. doi: 10.1177/0091270006292126. PMID 17101747
- [Result] Charlson ME, Carrozzino D, Guidi J, Patierno C. Charlson Comorbidity Index: A Critical Review of Clinimetric Properties. Psychother Psychosom. 2022;91(1):8-35. doi: 10.1159/000521288. Epub 2022 Jan 6. PMID 34991091
- [Result] Charlson ME, Pompei P, Ales KL, MacKenzie CR. A new method of classifying prognostic comorbidity in longitudinal studies: development and validation. J Chronic Dis. 1987;40(5):373-83. doi: 10.1016/0021-9681(87)90171-8. PMID 3558716
- [Result] Chougule PS, Najjar RP, Finkelstein MT, Kandiah N, Milea D. Light-Induced Pupillary Responses in Alzheimer's Disease. Front Neurol. 2019 Apr 12;10:360. doi: 10.3389/fneur.2019.00360. eCollection 2019. PMID 31031692
- [Result] de Vries L, Fouquaet I, Boets B, Naulaers G, Steyaert J. Autism spectrum disorder and pupillometry: A systematic review and meta-analysis. Neurosci Biobehav Rev. 2021 Jan;120:479-508. doi: 10.1016/j.neubiorev.2020.09.032. Epub 2020 Oct 22. PMID 33172600
- [Result] Detroyer E, Timmermans A, Segers D, Meyfroidt G, Dubois J, Van Assche A, Joosten E, Milisen K. Psychometric properties of the intensive care delirium screening checklist when used by bedside nurses in clinical practice: a prospective descriptive study. BMC Nurs. 2020 Apr 10;19:21. doi: 10.1186/s12912-020-00415-z. eCollection 2020. PMID 32308558
- [Result] Devlin JW, Skrobik Y, Gelinas C, Needham DM, Slooter AJC, Pandharipande PP, Watson PL, Weinhouse GL, Nunnally ME, Rochwerg B, Balas MC, van den Boogaard M, Bosma KJ, Brummel NE, Chanques G, Denehy L, Drouot X, Fraser GL, Harris JE, Joffe AM, Kho ME, Kress JP, Lanphere JA, McKinley S, Neufeld KJ, Pisani MA, Payen JF, Pun BT, Puntillo KA, Riker RR, Robinson BRH, Shehabi Y, Szumita PM, Winkelman C, Centofanti JE, Price C, Nikayin S, Misak CJ, Flood PD, Kiedrowski K, Alhazzani W. Clinical Practice Guidelines for the Prevention and Management of Pain, Agitation/Sedation, Delirium, Immobility, and Sleep Disruption in Adult Patients in the ICU. Crit Care Med. 2018 Sep;46(9):e825-e873. doi: 10.1097/CCM.0000000000003299. PMID 30113379
- [Result] Deyo RA, Cherkin DC, Ciol MA. Adapting a clinical comorbidity index for use with ICD-9-CM administrative databases. J Clin Epidemiol. 1992 Jun;45(6):613-9. doi: 10.1016/0895-4356(92)90133-8. PMID 1607900
- [Result] Ely EW, Inouye SK, Bernard GR, Gordon S, Francis J, May L, Truman B, Speroff T, Gautam S, Margolin R, Hart RP, Dittus R. Delirium in mechanically ventilated patients: validity and reliability of the confusion assessment method for the intensive care unit (CAM-ICU). JAMA. 2001 Dec 5;286(21):2703-10. doi: 10.1001/jama.286.21.2703. PMID 11730446
- [Result] Favre E, Bernini A, Morelli P, Pasquier J, Miroz JP, Abed-Maillard S, Ben-Hamouda N, Oddo M. Neuromonitoring of delirium with quantitative pupillometry in sedated mechanically ventilated critically ill patients. Crit Care. 2020 Feb 24;24(1):66. doi: 10.1186/s13054-020-2796-8. PMID 32093710
- [Result] Fiest KM, Soo A, Hee Lee C, Niven DJ, Ely EW, Doig CJ, Stelfox HT. Long-Term Outcomes in ICU Patients with Delirium: A Population-based Cohort Study. Am J Respir Crit Care Med. 2021 Aug 15;204(4):412-420. doi: 10.1164/rccm.202002-0320OC. PMID 33823122
- [Result] Gelinas C, Berube M, Chevrier A, Pun BT, Ely EW, Skrobik Y, Barr J. Delirium Assessment Tools for Use in Critically Ill Adults: A Psychometric Analysis and Systematic Review. Crit Care Nurse. 2018 Feb;38(1):38-49. doi: 10.4037/ccn2018633. PMID 29437077
- [Result] Gusmao-Flores D, Salluh JI, Chalhub RA, Quarantini LC. The confusion assessment method for the intensive care unit (CAM-ICU) and intensive care delirium screening checklist (ICDSC) for the diagnosis of delirium: a systematic review and meta-analysis of clinical studies. Crit Care. 2012 Jul 3;16(4):R115. doi: 10.1186/cc11407. PMID 22759376
- [Result] Hall CA, Chilcott RP. Eyeing up the Future of the Pupillary Light Reflex in Neurodiagnostics. Diagnostics (Basel). 2018 Mar 13;8(1):19. doi: 10.3390/diagnostics8010019. PMID 29534018
- [Result] Inouye SK. Delirium in older persons. N Engl J Med. 2006 Mar 16;354(11):1157-65. doi: 10.1056/NEJMra052321. No abstract available. PMID 16540616
- [Result] Inouye SK, Westendorp RG, Saczynski JS. Delirium in elderly people. Lancet. 2014 Mar 8;383(9920):911-22. doi: 10.1016/S0140-6736(13)60688-1. Epub 2013 Aug 28. PMID 23992774
- [Result] Jahns FP, Miroz JP, Messerer M, Daniel RT, Taccone FS, Eckert P, Oddo M. Quantitative pupillometry for the monitoring of intracranial hypertension in patients with severe traumatic brain injury. Crit Care. 2019 May 2;23(1):155. doi: 10.1186/s13054-019-2436-3. PMID 31046817
- [Result] Kim NY, Ryu SA, Kim YH. Factors Related to Delirium of Intensive Care Unit Patients in Korea: A Systematic Review. Iran J Public Health. 2021 Aug;50(8):1526-1535. doi: 10.18502/ijph.v50i8.6798. PMID 34917523
- [Result] Krewulak KD, Stelfox HT, Leigh JP, Ely EW, Fiest KM. Incidence and Prevalence of Delirium Subtypes in an Adult ICU: A Systematic Review and Meta-Analysis. Crit Care Med. 2018 Dec;46(12):2029-2035. doi: 10.1097/CCM.0000000000003402. PMID 30234569
- [Result] Maldonado JR. Delirium pathophysiology: An updated hypothesis of the etiology of acute brain failure. Int J Geriatr Psychiatry. 2018 Nov;33(11):1428-1457. doi: 10.1002/gps.4823. Epub 2017 Dec 26. PMID 29278283
- [Result] Nery RT, Reis AMM. Development of a Brazilian anticholinergic activity drug scale. Einstein (Sao Paulo). 2019 Apr 1;17(2):eAO4435. doi: 10.31744/einstein_journal/2019AO4435. PMID 30942279
- [Result] Oddo M, Taccone FS, Petrosino M, Badenes R, Blandino-Ortiz A, Bouzat P, Caricato A, Chesnut RM, Feyling AC, Ben-Hamouda N, Hemphill JC, Koehn J, Rasulo F, Suarez JI, Elli F, Vargiolu A, Rebora P, Galimberti S, Citerio G; ORANGE study investigators. The Neurological Pupil index for outcome prognostication in people with acute brain injury (ORANGE): a prospective, observational, multicentre cohort study. Lancet Neurol. 2023 Oct;22(10):925-933. doi: 10.1016/S1474-4422(23)00271-5. Epub 2023 Aug 28. PMID 37652068
- [Result] Okamoto S, Ishizawa M, Inoue S, Sakuramoto H. Use of Automated Infrared Pupillometry to Predict Delirium in the Intensive Care Unit: A Prospective Observational Study. SAGE Open Nurs. 2022 Sep 2;8:23779608221124417. doi: 10.1177/23779608221124417. eCollection 2022 Jan-Dec. PMID 36081493
- [Result] By the 2023 American Geriatrics Society Beers Criteria(R) Update Expert Panel. American Geriatrics Society 2023 updated AGS Beers Criteria(R) for potentially inappropriate medication use in older adults. J Am Geriatr Soc. 2023 Jul;71(7):2052-2081. doi: 10.1111/jgs.18372. Epub 2023 May 4. PMID 37139824
- [Result] Pisani MA, Murphy TE, Araujo KL, Slattum P, Van Ness PH, Inouye SK. Benzodiazepine and opioid use and the duration of intensive care unit delirium in an older population. Crit Care Med. 2009 Jan;37(1):177-83. doi: 10.1097/CCM.0b013e318192fcf9. PMID 19050611
- [Result] Reade MC. Is "behavioural disturbance" a clinically more useful concept than "delirium" for trials in intensive care medicine? Crit Care Resusc. 2023 Oct 18;23(2):125-127. doi: 10.51893/2021.2.ed1. eCollection 2021 Jun. No abstract available. PMID 38045519
- [Result] Riker RR, Sawyer ME, Fischman VG, May T, Lord C, Eldridge A, Seder DB. Neurological Pupil Index and Pupillary Light Reflex by Pupillometry Predict Outcome Early After Cardiac Arrest. Neurocrit Care. 2020 Feb;32(1):152-161. doi: 10.1007/s12028-019-00717-4. PMID 31069659
- [Result] Romano PS, Roos LL, Jollis JG. Adapting a clinical comorbidity index for use with ICD-9-CM administrative data: differing perspectives. J Clin Epidemiol. 1993 Oct;46(10):1075-9; discussion 1081-90. doi: 10.1016/0895-4356(93)90103-8. No abstract available. PMID 8410092
- [Result] Tune LE. Serum anticholinergic activity levels and delirium in the elderly. Semin Clin Neuropsychiatry. 2000 Apr;5(2):149-53. doi: 10.153/SCNP00500149. PMID 10837103
- [Result] van den Boogaard M, Pickkers P, Slooter AJ, Kuiper MA, Spronk PE, van der Voort PH, van der Hoeven JG, Donders R, van Achterberg T, Schoonhoven L. Development and validation of PRE-DELIRIC (PREdiction of DELIRium in ICu patients) delirium prediction model for intensive care patients: observational multicentre study. BMJ. 2012 Feb 9;344:e420. doi: 10.1136/bmj.e420. PMID 22323509
- [Result] van den Boogaard M, Schoonhoven L, Maseda E, Plowright C, Jones C, Luetz A, Sackey PV, Jorens PG, Aitken LM, van Haren FM, Donders R, van der Hoeven JG, Pickkers P. Recalibration of the delirium prediction model for ICU patients (PRE-DELIRIC): a multinational observational study. Intensive Care Med. 2014 Mar;40(3):361-9. doi: 10.1007/s00134-013-3202-7. Epub 2014 Jan 18. PMID 24441670
- [Result] Vasilevskis EE, Chandrasekhar R, Holtze CH, Graves J, Speroff T, Girard TD, Patel MB, Hughes CG, Cao A, Pandharipande PP, Ely EW. The Cost of ICU Delirium and Coma in the Intensive Care Unit Patient. Med Care. 2018 Oct;56(10):890-897. doi: 10.1097/MLR.0000000000000975. PMID 30179988
- [Result] Wassenaar A, Schoonhoven L, Devlin JW, van Haren FMP, Slooter AJC, Jorens PG, van der Jagt M, Simons KS, Egerod I, Burry LD, Beishuizen A, Matos J, Donders ART, Pickkers P, van den Boogaard M. Delirium prediction in the intensive care unit: comparison of two delirium prediction models. Crit Care. 2018 May 5;22(1):114. doi: 10.1186/s13054-018-2037-6. PMID 29728150
- [Result] Wilson JE, Mart MF, Cunningham C, Shehabi Y, Girard TD, MacLullich AMJ, Slooter AJC, Ely EW. Delirium. Nat Rev Dis Primers. 2020 Nov 12;6(1):90. doi: 10.1038/s41572-020-00223-4. PMID 33184265
- [Result] Wilson SF, Amling JK, Floyd SD, McNair ND. Determining interrater reliability of nurses' assessments of pupillary size and reaction. J Neurosci Nurs. 1988 Jun;20(3):189-92. doi: 10.1097/01376517-198806000-00011. PMID 2968419
- [Result] Wong HL, Weaver C, Marsh L, Mon KO, Dapito JM, Amin FR, Chauhan R, Mandal AKJ, Missouris CG. Polypharmacy and cumulative anticholinergic burden in older adults hospitalized with fall. Aging Med (Milton). 2023 Apr 5;6(2):116-123. doi: 10.1002/agm2.12250. eCollection 2023 Jun. PMID 37287675
- [Result] Yang E, Kreuzer M, Hesse S, Davari P, Lee SC, Garcia PS. Infrared pupillometry helps to detect and predict delirium in the post-anesthesia care unit. J Clin Monit Comput. 2018 Apr;32(2):359-368. doi: 10.1007/s10877-017-0009-z. Epub 2017 Mar 8. PMID 28275978
- [Result] Zhang M, Zhang X, Gao L, Yue J, Jiang X. Incidence, predictors and health outcomes of delirium in very old hospitalized patients: a prospective cohort study. BMC Geriatr. 2022 Mar 29;22(1):262. doi: 10.1186/s12877-022-02932-9. PMID 35351018